CLINICAL TRIAL: NCT01072825
Title: A European Network for the Investigation of Gender Incongruence
Acronym: ENIGI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2009/622
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Physical and Psychological Evaluation of Hormonal Therapy in Transsexual Persons
MeSH Terms: interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- transgender people starting hormone treatment
  Interventions: Other: questionnaires; Biological: blood sampling; Other: clinical evaluation; Other: Dermatology evaluation; Other: Bone evaluation

INTERVENTIONS:
Other: questionnaires — a descriptive questionnaire, SF-36, , bone questionnaires, Baecke physical activity questionnaire, voice evaluation
Biological: blood sampling — LFT (AST, ALT), CRP, creatinine, glucose, Total Cholesterol, Triglycerides, HDL-CH, LDL-CH, 25OH vitamin D, PSA if> 45 years, Hematocrit, testosterone, sex hormone-binding globulin, free testosterone , oestradiol, prolactin, luteinizing hormone, TSH, androgeengevoeligheids test (CAG RL), oral glucose tolerance test
Other: clinical evaluation — height, weight, blood pressure, chestcircumference, waist circumference, grip strength, measuring 2 ° and 4 ° finger, and Ferriman Gallwey score
Other: Dermatology evaluation — Evaluation of the hair pattern, using the Leeds acne classification scale, acne scars through ECCA scale (échelle d'évaluation clinique des cicatrices d'acné), androgenetic alopecia, and sebummetrie
Other: Bone evaluation — PQCT scanner, BMD assessment

SUMMARY:
The physical and psychological effects of the hormonal treatment of transsexual persons are not sufficiently described. 'Transparency' wants to answer this question in a prospective manner, in a multicenter study to describe these effects. The low prevalence of transsexualism was the stimulus to search for European partners for this Protocol. A common standardized hormonal protocol was designed.

ELIGIBILITY:
Inclusion Criteria:

* Transsexual persons older then 18 years, who are not yet treated with hormonal therapy.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: transsexual persons older than 18 years, who are not yet treated with hormonal therapy
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2010-02-15 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
physical and psychological effects of the hormonal treatment of transsexual persons | annually
  evaluations will be done every 3 months the first year of therapy, every 6 months in the second year, and after sex reassignment surgery annually.

CONTACTS AND LOCATIONS:
Overall Officials: Guy T'Sjoen, MD, Principal Investigator — University Hospital, Ghent
Locations (4):
- Genderteam UZ Gent, Ghent, Belgium
- Florence, Italy
- VU University Medical CenterAmsterdam, Amsterdam, Netherlands
- Rikshospitalet University Hospital, University of Oslo, Oslo, Norway

REFERENCES:
- [Derived] Shadid S, Abosi-Appeadu K, De Maertelaere AS, Defreyne J, Veldeman L, Holst JJ, Lapauw B, Vilsboll T, T'Sjoen G. Effects of Gender-Affirming Hormone Therapy on Insulin Sensitivity and Incretin Responses in Transgender People. Diabetes Care. 2020 Feb;43(2):411-417. doi: 10.2337/dc19-1061. Epub 2019 Nov 18. PMID 31740479
- [Derived] Auer MK, Ebert T, Pietzner M, Defreyne J, Fuss J, Stalla GK, T'Sjoen G. Effects of Sex Hormone Treatment on the Metabolic Syndrome in Transgender Individuals: Focus on Metabolic Cytokines. J Clin Endocrinol Metab. 2018 Feb 1;103(2):790-802. doi: 10.1210/jc.2017-01559. PMID 29216353
- [Derived] Bultynck C, Pas C, Defreyne J, Cosyns M, den Heijer M, T'Sjoen G. Self-perception of voice in transgender persons during cross-sex hormone therapy. Laryngoscope. 2017 Dec;127(12):2796-2804. doi: 10.1002/lary.26716. Epub 2017 Jul 21. PMID 28730692
- See also: website of the University Hospital of Ghent — http://www.uzgent.be